CLINICAL TRIAL: NCT06872658
Title: Exploratory Open-Label Study for the Development of a Method to Detect Dendritic Cell Recruitment in the Human Retina at Sites of Inflammatory Disease and Complement System Activation
Brief Title: Study to Detect Dendritic Cell Recruitment in Human Retina
Acronym: ICG-002
Status: Not yet recruiting | Type: Observational
Sponsor: MindImmune Therapeutics, Inc. (Industry)
Collaborators: Syneos Health (Other); CHU de Quebec-Universite Laval (Other)
Responsible Party: Sponsor
Other Study IDs: MindImmune
Record Dates: First submitted 2025-02-21; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-02

CONDITIONS: Dry Age Related Macular Degeneration; Mild Cognitive Impairment (MCI); Alzheimer Disease
Keywords: AMD; Dry Age Related Macular Degeneration; AD; MCI; Mild Cognitive Impairment; Alzheimer Disease
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Participants with Dry AMD with GA: To determine if human phagocytic cells labeled with the near-infrared dye ICG in the periphery can subsequently be detected in association with retinal pathology in patients with Dry AMD with geographic atrophy (GA).
- Healthy Older Adult Participants: To determine if human phagocytic cells labeled with the near-infrared dye ICG in the periphery can subsequently be detected in association with retinal pathology in healthy elderly patients
- Participants with Mild Cognitive Impairment (MCI) due to AD or mild AD: To determine if human phagocytic cells labeled with the near-infrared dye ICG in the periphery can subsequently be detected in association with retinal pathology in patients patients diagnosed with either mild cognitive impairment (MCI) due to Alzheimer's disease (AD

SUMMARY:
The goal of this study is to develop an optimal method to detect the immune cells (cells that protect the human body against diseases) in association with abnormal conditions of the retina (light sensitive tissue in the back of the eye) that will be relevant to diseases such as age related macular degeneration (AMD), mild cognitive impairment (MCI) due to Alzheimer's Disease (AD) or mild AD.

The main objectives of this study are:

1. Establish Optimal Method for Retinal Imaging of Dendritic Cells (DCs)
2. Safety and Tolerability of ICG infusion in normal healthy, older adult volunteers, in participants with AMD (Dry AMD with Geographic Atrophy (GA)), and in participants who have received a diagnosis of either Mild Cognitive Impairment (MCI) due to AD, or mild AD

DETAILED DESCRIPTION:
This methods development pilot study is intended to determine if human phagocytic cells labeled with the near-infrared dye ICG in the periphery can subsequently be detected in association with retinal pathology in two cohorts of participants: 1) patients with Dry AMD with geographic atrophy (GA), N = 2-6; and 2) patients diagnosed with either mild cognitive impairment (MCI) due to Alzheimer's disease (AD) or with mild AD, N = 2-6. Conversely, it is hypothesized that these cells will be largely absent in healthy control participants (N = 2-3). For both disease conditions, retinal pathology includes inclusions that contain amyloid plaques, areas of retinal thinning and neuronal loss, damage to the RPE and choroid, and changes in vascular structure. Accumulation of ICG-labeled cells should be seen close to the border(s) of GA in the Dry AMD participants. The imaging results for each participant will be reviewed by the study team to modify the imaging approach for the next participant. A maximum of fifteen (15) subjects will be recruited for participation, and a maximum of 3 of these participants will be healthy control participants without any retinal pathology.

ELIGIBILITY:
Inclusion Criteria:

1. All Study Participants

   * Male or female and between the ages of 55 to 80 years old (inclusive)
   * Participants are determined by the qualified investigator to be medically stable and able to understand and agree to comply with the study procedures and report for scheduled study visits.
   * Participants have adequate hearing, vision, and language skills to provide informed consent and to cooperate with all retinal imaging, cognitive testing, interviews and other medical procedures as specified in the protocol. Hearing augmentation (i.e., hearing aids) are allowed.
   * Participants are able to reliably communicate with study personnel about adverse events (AEs) and concomitant medications.
   * Provide signed written informed consent according to institutional guidelines. Participants with mild AD must be able to provide assent and be accompanied by a relative or caregiver who is empowered to provide written consent.
   * Permitted medications stable for at least 1 month prior to screening. In particular:

     * Participants may take stable doses of antidepressants lacking significant anticholinergic side effects (if they are not currently depressed and do not have a history of major depression within the past year).
2. Healthy Elderly Participants

   * MMSE score > 27
   * CDR score = 0
   * No current or past history of first-degree relative(s) with either a diagnosis of AD or suspected AD, and no subjective memory impairment with persisting worries.
   * If any such test results are available, no APOE e4 allele positivity or abnormal beta-amyloid protein aggregation as assessed by blood plasma, PET imaging or CSF analyses.
   * No evidence of any retinal/ocular diseases, other than myopia or hyperopia
   * No evidence of any neurological / neurodegenerative diseases
3. Participants with Dry AMD with GA

   * MMSE score > 27
   * CDR score = 0
   * Advanced non-neovascular stage AMD, as determined by qualified neuro-ophthalmologist or retinal specialist
   * No evidence of choroidal neovascularization (CNV) in study eye - current or historical
   * Best Corrected Visual Acuity (BCVA) ≥ 20/80
   * Low-luminance visual acuity deficit, defined as the difference between BCVA and LLVA > 5 letters
   * Cumulative GA lesion size 1.27 mm2 (approximately ≥ 0.5 disc area (DA)) and ≤ 10.16 mm2 (approximately ≤ 4.0 DA). Standard DA is equivalent to 2.54 mm2 on the retina.
   * Participants with Dry AMD who are not (yet) being treated with a complement system inhibitor (intravitreal injections).
4. Participants with Mild Cognitive Impairment (MCI) due to AD or mild AD

   * MMSE score > 21
   * CDR score between 0.5 and 1.0
   * MoCA total score > 18 and < 26 at screening
   * Positive prior biomarker evidence of Alzheimer's disease (blood plasma marker(s), PET imaging, or CSF assays), by review of available medical records
   * A clinical diagnosis of either mild cognitive impairment (MCI) due to AD, or mild AD, from qualified specialist or from a memory disorders clinic or center
   * Participants must have a study partner (i.e., family member, close friend, or caregiver) who can attend study appointments with them.
   * Because this study does not include any form of therapeutic intervention, participants' concurrent enrollment in other clinical trials for MCI or AD is allowed, including those that involved the use of investigational drugs. Relevant information about other studies in which individuals are participating (e.g., study name, sponsor) will be made available and recorded on their case report forms (CRFs).

Exclusion Criteria:

1. Medical History

   * Participants with a history of any anaphylactic reactions to drugs
   * Participants with a history of allergic reaction to ICG
   * Participants with a history of iodine sensitivity and/or allergic reaction to iodine
   * Participants with a history of a clinically significant hepatic disease
   * Participants with a Modified Hachinski Ischemia Scale (MHIS) score > 2
   * Participants with a known hypersensitivity to tropicamide eye drops or other anticholinergic medications
2. Participants with histories of other ocular or neurologic disease that could affect the results including, but not limited to, diabetic retinopathy or glaucoma.
3. Geriatric Depression Scale Short Form (GDS-S 15 Items) score > 6.
4. Target Disease Exceptions

   * Any participant diagnosed to have an autoimmune disorder, including but not limited to

     * Psoriasis
     * Lupus
     * Rheumatoid arthritis
     * Crohn's disease
     * Multiple sclerosis
     * Alopecia areata
   * Any participant who has any unstable cardiovascular (included uncontrolled hypertension), pulmonary, or GI disease.
   * History of alcohol or substance abuse and/or dependence within the past 2 years (DSM-V criteria).
   * History of schizophrenia or a history of psychotic features, agitation or behavioral problems within the last 3 months, which could lead to difficulty complying with the protocol.
   * Participants who, in the investigator's opinion, will not comply with study procedures.
   * Participants who, in the investigator's opinion, have any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including (but not limited to):

     * History of myocardial infarction within the past six (6) months or unstable or severe cardiovascular disease including angina or CHF with symptoms at rest.
     * Uncontrolled hypertension (i.e., systolic BP > 170 or diastolic BP > 100)
     * Uncontrolled (A1C>7) or insulin requiring diabetes.
     * History of symptoms of narrow-angle glaucoma (warning signs include eye pain, restricted vision, blurred vision)
     * History of elevated intraocular pressure, or medical record evidence of intraocular pressure > 20 mm Hg
5. Concurrent Medications

   * Any participant who is immunocompromised at screening including taking medications that are systemic immunosuppressives including corticosteroids but not NSAIDS
   * Any participant currently prescribed a biologic immunosuppressive therapy or having taken such therapy in the prior 3 months, including

     * abatacept (Orencia)
     * adalimumab (Humira)
     * anakinra (Kineret)
     * certolizumab (Cimzia)
     * etanercept (Enbrel)
     * golimumab (Simponi)
     * infliximab (Remicade)
     * ixekizumab (Taltz)
     * natalizumab (Tysabri)
     * rituximab (Rituxan)
     * secukinumab (Cosentyx)
     * tocilizumab (Actemra)
     * ustekinumab (Stelara)
     * vedolizumab (Entyvio)
     * Monoclonal antibodies
     * basiliximab (Simulect)
     * daclizumab (Zinbryta)
   * Regular (daily) use of narcotics or antipsychotic medications. Low doses for off-label use may be permitted, as determined by the principal investigator's clinical judgment and if stable for 4 weeks prior to screening.
   * New use of anti-Parkinsonian medications (e.g., sinemet, amantaine, bromocriptine, pergolide and selegiline) within 2 months prior to screening. Low doses for off-label use may be permitted, as determined by the principal investigator's clinical judgment and if stable for 2 months prior to screening.
   * New use of anti-convulsants (e.g., phenytoin, phenobarbital, carbamazepine) within 2 months prior to screening. Low doses for off-label use may be permitted, as determined by the principal investigator's clinical judgment and if stable for 2 months prior to screening.
   * New use of centrally active beta-blockers, narcotics, methyldopa and clonidine within 4 weeks prior to screening.
   * New use of neuroleptics or narcotic analgesics within 4 weeks prior to screening.
   * New and chronic use of long-acting benzodiazepines or barbiturates within 4 weeks prior to screening.
   * Initiation or change in dose of an antidepressant within 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable)
   * Any participant currently or previously treated for Dry AMD with a complement system inhibitor.
6. Physical and Laboratory Test Findings at Screening

   * Any participant, in the clinical judgement of the qualified investigator, with uncontrolled hypertension, abnormal systolic BP, or abnormal heart rate at screening (e.g., repeated diastolic measurements ≥ 96 mmHg).
   * Any participant with either of the following hepatic test abnormalities at screening:

     * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.0 times the institutional ULN
     * Total Bilirubin > 2 times the institutional ULN
   * Any participant with P-Amylase or Lipase values > 2 times the ULN at screening
   * Any participant at screening with insulin-dependent diabetes mellitus or HbA1C ≥ 6.5%
   * Abnormal liver function test laboratory results, as determined by screening visit (pre-ICG infusion) safety lab tests
   * Any participant at screening with pathologic renal findings as defined by the presence of calculated glomerular filtration rate (GFR) (creatinine clearance) ≤45 ml/min/1.73m2 (2021 revision of CKD-EPI formula for GFR estimate)
   * Any participant at screening with any of the following hematologic abnormalities:

     * Hemoglobin < 10g/dL
     * WBC < 3.0 x 103/mm3
     * Platelet count < 100,000/mm3
   * Any participant who has a known infection with a human immunodeficiency virus, hepatitis B virus, or hepatitis C virus.
   * Any participant with a positive urine drug screen with no concomitant medication to justify the results.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Between 2 and 15 participants, as needed to establish methods. Between one (1) and (3) of these participants will be healthy control participants without any retinal pathology. Up to six (6) Dry AMD with GA participants and up to six (6) MCI and/or mild AD participants will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Determining Method to detect ICG immune cells both AMD and AD Patients | Retinal Scans are completed 30 minutes prior to start of ICG infusion (Baseline),240 and 360 minutes after start of ICG infusion. Each retinal scan takes 12-15 minutes.
  Detecting ICG-labeled immune cells in association with retinal pathology that will be relevant to Age-Related Macular Degeneration (AMD) and to Alzheimer's disease (AD).
Establish duration and dosage of ICG infusion | Retinal Scans are completed 30 minutes prior to start of ICG infusion (Baseline),240 and 360 minutes after start of ICG infusion. Each retinal scan takes 12-15 minutes.
  Set duration and dosage of ICG infusion to optimize resolution of Dendritic Cells with fundus autofluorescence (FAF) imaging and/or ICG fluoroscopy.
Establish time intervals between ICG dosing and retinal imaging | Retinal Scans are completed 30 minutes prior to start of ICG infusion (Baseline),240 and 360 minutes after start of ICG infusion. Each retinal scan takes 12-15 minutes.
  Determine optimal time interval(s) between ICG infusion and retinal imaging to identify labeled Dendritic Cells.
Verify locations of Dendritic Cells | Retinal Scans are completed 30 minutes prior to start of ICG infusion (Baseline),240 and 360 minutes after start of ICG infusion. Each retinal scan takes 12-15 minutes.
  Verify location of DCs by utilizing 3D retinal SD-OCT and FAF imaging.
Safety data analyses will be conducted on all subjects who have started the infusion of ICG | Safety and Tolerability measures are assessed beginning from the signing of the ICF through the End of study (Telephone Follow-up Days 8-15).
  The number and percentage of participants experiencing 1 or more AEs will be summarized by participant group, relationship to Test Product administration, and severity. AEs will be coded using Medical Dictionary for Regulatory Activities (MedDRA) terminology. Listings of participants who withdraw from the study due to an AE, serious AEs and/or death will be presented. Laboratory parameters will be summarized for each cohort using descriptive statistics and data listings of clinically significant abnormalities. Vital signs and ECG data will be summarized by changes from baseline values using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Syder, PhD, Study Director — MindImmue

IPD SHARING:
Plan to Share IPD: No